CLINICAL TRIAL: NCT00886561
Title: HIV- Risk Reduction Behavioral Intervention for Commercial Sex Workers in Yerevan Armenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: American University of Armenia (Other)
Responsible Party: Principal Investigator, Ralph J. DiClemente, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0126-2005; ARX1-2719-YE-06 (Other: Other)
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: HIV Prevention; HIV Infections
Keywords: HIV prevention, female sex workers; HIV seronegativity
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIV risk reduction intervention (Experimental): Behavioral intervention designed to reduce HIV risk behaviors and enhance enhance HIV-preventive behaviors among female sex workers (FSWs) in Armenia
  Interventions: Behavioral: HIV risk reduction intervention
- Wait list control (Active Comparator): Will receive behavioral intervention after completion of study upon request.
  Interventions: Behavioral: HIV risk reduction intervention

INTERVENTIONS:
Behavioral: HIV risk reduction intervention — Education intervention designed to reduce HIV risk behaviors and enhance HIV prevention behaviors among female sex workers in Armenia

SUMMARY:
This pilot study will test the efficacy of a behavioral intervention in reducing HIV related risk behaviors among sex workers in Yerevan, Armenia.

DETAILED DESCRIPTION:
The purpose of this pilot study is to evaluate the efficacy of an intervention to reduce sexual risk behaviors and enhance HIV-preventive behaviors among female sex workers (FSWs) in Yerevan, Armenia. The study design is a randomized controlled trial of 120 FSWs aged 18 and over recruited through Hope and Help NGO. Participants will complete an interviewer administered questionnaire collected at baseline, 3- and 6-month follow-up.

Subsequently, participants will be randomly assigned to either the intervention condition or a wait-list control. Those randomized to the intervention condition will receive a 2-hour one-on-one intervention session emphasizing HIV knowledge, self-efficacy, and condom use behaviors. They will also receive a 10-15 minute booster session at 3-month follow-up. The comparison condition is wait-listed, but have the choice of participating in the intervention program upon completion of the study.

The main outcome measure includes consistent condom use, defined as condom use during every episode of vaginal intercourse with clients. Other outcome measures are condom application by FSW and HIV- preventive behaviors such as condom use self-efficacy, knowledge of HIV transmission dynamics,perceived barriers to condom use and condom use errors.

Results from this pilot study are expected to inform a larger trial to be implemented with FSWs in Armenia, in an effort to devise gender and culturally relevant intervention programs to prevent HIV transmission in this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* traded sex for money in the past 7 days
* cognitive ability to participate in assessment and intervention

Exclusion Criteria:

* younger than 18 years of age
* did not trade sex for money in the past 7 days
* cognitively unable to participate in assessment and intervention

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-07; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Consistent condom use | 3 and 6 months post intervention

SECONDARY OUTCOMES:
Condom application | 3 and 6 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ralph J DiClemente, PhD, Principal Investigator — Emory University
Locations (1):
- Hope and Help NGO, Yerevan, Yerevan, Armenia